CLINICAL TRIAL: NCT07076225
Title: A Ultrashort Regimen for Drug-susceptible Pulmonary Tuberculosis in Elderly Patients: A Multicenter Randomized Controlled Trial
Brief Title: Ultra-Short Regimen for Elderly DS-TB
Acronym: Elderly-USR
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Shenzhen Third People's Hospital (Other)
Collaborators: Beijing Chest Hospital, Capital Medical University (Other); Fudan University (Other); West China Hospital (Other); Huazhong University of Science and Technology (Other); Tsinghua University (Other)
Responsible Party: Principal Investigator, Shuihua Lu, Professor, Shenzhen Third People's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USRElderly
Record Dates: First submitted 2025-06-30; First posted 2025-07-22 (Actual); Last update posted 2025-07-22 (Actual); Status verified 2025-07

CONDITIONS: Pulmonary Tuberculosis
MeSH Terms: conditions — Tuberculosis, Pulmonary | interventions — bedaquiline; sitafloxacin; Linezolid; Pyrazinamide; Isoniazid; Protons; Rifampin; Ethambutol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Drug-susceptible TB (A) (Experimental): 2 months (9 weeks) BLSZ regimen: The treatment involves the use of bedaquiline (B), linezolid (L), sitafloxacin (S), and pyrazinamide (Z) throughout the entire process. At the end of 2 months (9 weeks) of treatment, if the sputum smear is still positive or if clinical symptoms have not improved, the treatment duration can be extended to 13 weeks. After the extended treatment period (3 months or 13 weeks), if the sputum smear remains positive or if clinical symptoms have not been relieved, the patient should be switched to the standard treatment regimen, and the subject should be withdrawn from the study.
  Interventions: Drug: Bedaquiline (B); Drug: Sitafloxacin (S); Drug: Linezolid (L); Drug: Pyrazinamide (Z)
- Drug-susceptible TB (B) (Active Comparator): 2HRZE/4HR (26 weeks): Four drugs-isoniazid (H), rifampicin (R), pyrazinamide (Z), and ethambutol (E)-are used during the first 2 months of the intensive phase. This is followed by 4 months of consolidation treatment, during which only isoniazid and rifampicin are used.
  Interventions: Drug: Pyrazinamide (Z); Drug: Isoniazid (H); Drug: Rifampicin (R); Drug: Ethambutol (E)

INTERVENTIONS:
Drug: Bedaquiline (B) — The initial dose of bedaquiline is 400 mg daily for 2 weeks, followed by 200 mg three times a week.
  Arms: Drug-susceptible TB (A)
Drug: Sitafloxacin (S) — 200mg once daily
  Arms: Drug-susceptible TB (A)
Drug: Linezolid (L) — 600mg once daily
  Arms: Drug-susceptible TB (A)
Drug: Pyrazinamide (Z) — 20-30 mg/kg/day; 1000 mg for patients weighing <50 kg, 1500 mg for patients weighing ≥50 kg but <75 kg, and 2000 mg for patients weighing ≥75 kg.
Drug: Isoniazid (H) — 4-6 mg/kg once daily, 300 mg once daily
  Arms: Drug-susceptible TB (B)
Drug: Rifampicin (R) — 8-12 mg/kg once daily, 450 mg for patients weighing <50 kg, 600 mg for patients weighing ≥50 kg but <75 kg, and 750 mg for patients weighing ≥75 kg.
  Arms: Drug-susceptible TB (B)
Drug: Ethambutol (E) — 15-25 mg/kg once daily, 750 mg once daily
  Arms: Drug-susceptible TB (B)

SUMMARY:
Tuberculosis (TB) remains one of the leading global public health concerns and is among the top ten causes of death from a single infectious agent. China ranks third worldwide in total TB burden, with a substantial proportion of cases classified as drug-susceptible TB (DS-TB). Despite the availability of effective standard treatment regimens, the current 6-month therapy duration poses challenges in terms of patient adherence, resource allocation, and overall treatment success.

In recent years, ultrashort-course regimens for DS-TB have been proposed and evaluated in clinical studies, showing promising results in improving adherence, reducing treatment duration, and maintaining or even enhancing treatment efficacy. However, these regimens have primarily been studied in younger populations, with limited data available for elderly patients. Older adults often present with age-related physiological changes, multiple comorbidities, and an increased risk of adverse drug reactions, which may affect both the efficacy and safety of treatment.

Therefore, this study aims to assess the therapeutic effectiveness and safety profile of a novel ultrashort-course regimen for drug-susceptible pulmonary TB specifically in patients aged 65 years and older.

ELIGIBILITY:
Inclusion criteria:

1. Aged 65 years or older, regardless of gender
2. Clinical symptoms and/or pulmonary imaging (chest X-ray or chest CT) support the diagnosis of active pulmonary tuberculosis;
3. Microbiological testing (molecular or phenotypic) confirms the presence of Mycobacterium tuberculosis, and susceptible to rifampicin; Recommend using respiratory specimens for GeneXpert MTB/RIF testing;
4. Voluntarily sign the informed consent form for participating in this project and be able and willing to accept follow-up visits;
5. Willing to undergo HIV testing;
6. Willing to preserve samples including DNA;

Exclusion criteria:

1. Prior to this study, patients who were diagnosed with active pulmonary tuberculosis and had received anti-tuberculosis treatment (including first-line and second-line anti-tuberculosis drugs);
2. Intolerance or allergy to any investigational drug (i.e., bedaquiline, linezolid, pyrazinamide, etc);
3. Resistance to any investigational drug (i.e., bedaquiline, linezolid, pyrazinamide, etc). The following detection methods can be used: tNGS or other drug sensitivity testing methods (such as GeneXpert MTB/XDR, dissolution curve method, phenotypic drug sensitivity, etc.);
4. Suffering from hematogenous disseminated tuberculosis or coexisting with extrapulmonary tuberculosis (as specified in this study, the scope of pulmonary tuberculosis includes: simple pulmonary tuberculosis, pulmonary tuberculosis + tuberculous pleurisy/bronchial tuberculosis/mediastinal lymph node tuberculosis. Extrapulmonary tuberculosis refers to tuberculosis other than the chest-related types mentioned above);
5. Presence of non-tuberculous mycobacteria or other microbial lung infections that affect treatment outcomes;
6. Simultaneously using drugs that affect the efficacy of this study or have contraindications for combination therapy;
7. Use of any immunosuppressive medication or systemic glucocorticoids for more than 2 weeks before screening;
8. Any medication currently used or planned to be used that is known to significantly prolong the QTc interval, including but not limited to: amiodarone, amitriptyline, chloroquine, chlorpromazine, cisapride, dipyridamole, itraconazole, procaine, quinidine, or sotalol;
9. Uncontrolled blood sugar in diabetes, with no likelihood of improving blood sugar status according to the judgment of the researchers;
10. HIV positive;
11. Coexisting with severe autoimmune diseases, severe liver and kidney dysfunction, psychiatric disorders, hematological disorders, or malignant tumors;
12. Laboratory parameters within 14 days prior to recruitment: (1) Serum AST and ALT levels ≥ 3 times the upper limit of normal (ULN); (2) Blood creatinine ≥ 2 times ULN; (3) Hemoglobin ≤ 70 g/L; (4) Platelet count ≤ 50 × 10^9/L; (5) Blood potassium levels are ≥ 5.5 mmol/L or ≤ 3.5 mmol/L;
13. ECG QTcF ≥450 ms (allowing for one re-test during the screening phase to reassess eligibility for inclusion); Presence of one or more risk factors that could cause QT interval prolongation, such as arrhythmia, myocardial ischemia, etc.; history or family history of long QT syndrome;
14. Weight <30 kg, or ≥90 kg;
15. The patient has participated in clinical trials of other drugs within the past 3 months during the screening period;
16. Other conditions deemed unsuitable for participation in the study by the research doctors.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2025-07-25 (Estimated); Primary Completion 2030-01-31 (Estimated); Study Completion 2030-07-31 (Estimated)

PRIMARY OUTCOMES:
Unfavorable outcomes | 12 months (52 weeks)
  Percentage of patients with unfavorable outcomes (failure, treatment interruption, death, loss to follow-up, re-treatment, recurrence) at 12 months (52 weeks) after randomization
Percentage of patients with treatment interruption | 2 months (9 weeks)
  Percentage of patients who have treatment interruption due to any reason （including death）within 2 months (9 weeks) after randomization

SECONDARY OUTCOMES:
Sputum culture conversion rate | 2 months (9 weeks) after randomization
Serious adverse events or grade 3 or higher adverse events (short-term) | 12 months (52 weeks) after randomization
Serious adverse events or grade 3 or higher adverse events (mid-term) | 18 months (78 weeks) after randomization
Adverse events during treatment | 26 weeks
Percentage of patients with QTcF prolongation | 26 weeks
Percentage of Patients with liver function damage | 26 weeks

REFERENCES:
- [Background] Paton NI, Cousins C, Suresh C, Burhan E, Chew KL, Dalay VB, Lu Q, Kusmiati T, Balanag VM, Lee SL, Ruslami R, Pokharkar Y, Djaharuddin I, Sugiri JJR, Veto RS, Sekaggya-Wiltshire C, Avihingsanon A, Sarin R, Papineni P, Nunn AJ, Crook AM; TRUNCATE-TB Trial Team. Treatment Strategy for Rifampin-Susceptible Tuberculosis. N Engl J Med. 2023 Mar 9;388(10):873-887. doi: 10.1056/NEJMoa2212537. Epub 2023 Feb 20. PMID 36808186